CLINICAL TRIAL: NCT03399500
Title: m-Health to Increase Service Utilization in Recently Incarcerated Homeless Adults
Brief Title: Homeless Care Management App
Acronym: Link2Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: The University of Texas Health Science Center, Houston (Other); National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8525; HSC-SPH-15-0632 (Other: UTHealth IRB); 1R01MD010733-01A1 (NIH)
Record Dates: First submitted 2017-12-22; First posted 2018-01-16 (Actual); Results first posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Substance Use Disorders; Mental Health Impairment; Health Behavior; Adherence, Patient
Keywords: Case Management; Homelessness; Smartphone; Health Related Quality of Life; Mental Health; Substance Use Disorders
MeSH Terms: conditions — Substance-Related Disorders; Health Behavior; Patient Compliance; Psychological Well-Being | interventions — Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Case Management (UCM) (Active Comparator): Group receives standard case management at the shelter
  Interventions: Behavioral: In-Person Case Management at Homeless Recovery Program
- UCM + Smartphone (Experimental): Group receives standard case management and an unlimited smartphone
  Interventions: Behavioral: In-Person Case Management at Homeless Recovery Program; Behavioral: Unlimited Smartphone
- Smartphone Based Case Management (SPCM) (Experimental): Group receives standard case management and an unlimited smartphone with the SPCM app
  Interventions: Behavioral: In-Person Case Management at Homeless Recovery Program; Behavioral: Unlimited Smartphone; Behavioral: Smartphone Based Case Management (SPCM) app

INTERVENTIONS:
Behavioral: In-Person Case Management at Homeless Recovery Program — In-Person Case Management at Homeless Recovery Program
Behavioral: Unlimited Smartphone — Smartphone with unlimited calls, texts, and data plan
  Arms: Smartphone Based Case Management (SPCM); UCM + Smartphone
Behavioral: Smartphone Based Case Management (SPCM) app — Smartphone Based Case Management app
  Arms: Smartphone Based Case Management (SPCM)

SUMMARY:
There is a significant revolving door of incarceration among homeless adults, a population with substantial health disparities. Homeless adults who receive the professional coordination of individualized care (i.e., case management) during the period following their release from jail experience fewer mental health and substance use problems, are more likely to obtain stable housing, and are less likely to be re-incarcerated. The proposed study will use mobile technology to address these barriers and fill gaps in the understanding of the causes of the revolving door of homeless incarceration. This research represents a step toward integrated service connection and healthcare service provision for one of the most underserved, high need, and understudied populations in the United States. Smart phone apps that increase the use of available healthcare services and identify predictors of key outcomes (e.g., homelessness, re-arrest, medication compliance) could be used to reach hard to reach populations with histories of significant and persistent health disparities (e.g., homeless adults).

ELIGIBILITY:
Inclusion Criteria:

* released from Dallas County Jail in the past month
* plan to reside in the Dallas area for the next year
* enrolled in The Bridge Homeless Recovery Program
* willing and able to attend the baseline visit, randomization visit, and the 1, 3, and 6-month follow-up visits
* score ≥ 4 on the REALM-SF indicating > 6th grade English literacy level
* score >24 on the Mini-Mental State Exam indicating no substantial cognitive impairment.

Exclusion Criteria

* Cannot read English
* Under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Businelle, Ph.D., Principal Investigator — University of Oklahoma; Jennifer M Reingle, Ph.D., Principal Investigator — UTHealth School of Public Health
Locations (2):
- United States (2):
  - University of Oklahoma Health Sciences Center - OTRC, Oklahoma City, Oklahoma
  - UTHealth School of Public Health, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reingle Gonzalez JM, Businelle MS, Kendzor D, Staton M, North CS, Swartz M. Using mHealth to Increase Treatment Utilization Among Recently Incarcerated Homeless Adults (Link2Care): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2018 Jun 5;7(6):e151. doi: 10.2196/resprot.9868. PMID 29871852

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Case Management (UCM) | UCM + Smartphone | Smartphone Based Case Management (SPCM)
Started | 136 | 134 | 133
Completed | 64 | 72 | 81
Not Completed | 72 | 62 | 52

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Case Management (UCM) | UCM + Smartphone | Smartphone Based Case Management (SPCM) | Total
Number analyzed (Participants) | 136 | 134 | 133 | 403
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.68 (10.63) | 40.88 (11.37) | 40.46 (10.84) | 40.34 (10.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 19 | 56
  Male | 118 | 115 | 114 | 347
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 17 | 17 | 51
  Not Hispanic or Latino | 119 | 117 | 116 | 352
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 2 | 7
  Asian | 1 | 1 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 86 | 87 | 67 | 240
  White | 33 | 29 | 32 | 94
  More than one race | 11 | 10 | 19 | 40
  Unknown or Not Reported | 2 | 5 | 11 | 18
Region of Enrollment [Number; unit: participants]
  United States | 136 | 134 | 133 | 403

OUTCOME MEASURES:

1. Primary Outcome: Number of Case Management Sessions Completed
Description: Total number of sessions completed between the randomization visit and 6-month follow-up
Time Frame: 6-month follow-up
Measure: Mean (Standard Deviation); unit: number of sessions
Arm/Group | Usual Case Management (UCM) | UCM + Smartphone | Smartphone Based Case Management (SPCM)
Number analyzed (Participants) | 136 | 134 | 133
number of sessions | 9.39 (11.40) | 7.69 (10.79) | 8.46 (11.17)

2. Secondary Outcome: Number of Homeless Nights
Description: Total number of self-reported homeless nights over the 6 month study period (via Timeline Follow Back Procedures). Participants with any missing are excluded.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: number of nights
Arm/Group | Usual Case Management (UCM) | UCM + Smartphone | Smartphone Based Case Management (SPCM)
Number analyzed (Participants) | 46 | 56 | 61
number of nights | 161.48 (41.64) | 167.12 (31.19) | 159.00 (39.09)

3. Secondary Outcome: Number of Re-arrests
Description: Total number of times each participant is booked into Dallas County Jail (using jail arrest records)
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: number of arrests
Arm/Group | Usual Case Management (UCM) | UCM + Smartphone | Smartphone Based Case Management (SPCM)
Number analyzed (Participants) | 136 | 134 | 133
number of arrests | 0.55 (0.82) | 0.64 (1.01) | 0.61 (1.06)

4. Secondary Outcome: Alcohol Use
Description: Number of days of alcohol use (via Timeline Follow Back procedures). Any participant that missed any of the follow-ups are missing.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Usual Case Management (UCM) | UCM + Smartphone | Smartphone Based Case Management (SPCM)
Number analyzed (Participants) | 46 | 56 | 61
days | 14.26 (31.93) | 20.70 (39.09) | 26.57 (41.37)

5. Secondary Outcome: Drug Use
Description: Number of days of drug use (via Timeline Follow Back procedures). Any participant that missed any of the 3 follow-ups are missing.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Usual Case Management (UCM) | UCM + Smartphone | Smartphone Based Case Management (SPCM)
Number analyzed (Participants) | 46 | 56 | 61
days | 6.33 (16.75) | 22.34 (48.32) | 17.61 (32.64)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Definition does not differ from the clinicaltrials.gov definitions.
Arm/Group | Usual Case Management (UCM) | UCM + Smartphone | Smartphone Based Case Management (SPCM)
All-Cause Mortality (participants affected / at risk) | 0/136 | 0/134 | 0/133
Serious Adverse Events (participants affected / at risk) | 0/136 | 0/134 | 0/133
Other Adverse Events (participants affected / at risk) | 0/136 | 0/134 | 0/133

LIMITATIONS AND CAVEATS:
There are no limitations or caveats to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/00/NCT03399500/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/00/NCT03399500/ICF_001.pdf